CLINICAL TRIAL: NCT03922048
Title: A Phase 2, 2-Part, Open-Label, Dose-Finding and Double-Blind Study to Assess the Pharmacokinetics, Pharmacodynamics, and Safety of HTX-011 for Postoperative Analgesia in Adolescents and Children (≥3 to <17 Years of Age) Undergoing Unilateral Open Inguinal Herniorrhaphy
Brief Title: Pediatric Postoperative Analgesia Herniorrhaphy Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to lack of enrollment.
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: HTX-011-216
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Analgesia
Keywords: inguinal hernia; postoperative pain; herniorrhaphy; pediatric; local anesthetic
MeSH Terms: conditions — Agnosia; Hernia, Inguinal; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (10):
- Cohort 1 Part A: HTX-011 (Experimental): Adolescents ≥12 to <17 years of age. A single dose of HTX-011 via instillation into the surgical site.
  Interventions: Drug: HTX-011; Device: Luer Lock Applicator
- Cohort 1 Part A: bupivacaine HCl (Active Comparator): Adolescents ≥12 to <17 years of age. A single dose of bupivacaine HCl 0.25% (without epinephrine) via injection into the surgical site.
  Interventions: Drug: Bupivacaine HCl
- Cohort 1 Part B: HTX-011 (Experimental): Adolescents ≥12 to <17 years of age. Dose to be determined from Cohort 1 Part A.
  Interventions: Drug: HTX-011; Device: Luer Lock Applicator
- Cohort 1 Part B: bupivacaine HCl (Active Comparator): Adolescents ≥12 to <17 years of age. A single dose of bupivacaine HCl 0.25% (without epinephrine) via injection into the surgical site
  Interventions: Drug: Bupivacaine HCl
- Cohort 2 Part A: HTX-011 (Experimental): Children ≥6 to <12 years of age. Dose to be determined from Cohort 1.
  Interventions: Drug: HTX-011; Device: Luer Lock Applicator
- Cohort 2 Part A: bupivacaine HCl (Active Comparator): Children ≥6 to <12 years of age. A single dose of bupivacaine HCl 0.25% (without epinephrine) via injection into the surgical site
  Interventions: Drug: Bupivacaine HCl
- Cohort 2 Part B: HTX-011 (Experimental): Children ≥6 to <12 years of age. Dose to be determined from Cohort 1.
  Interventions: Drug: HTX-011; Device: Luer Lock Applicator
- Cohort 2 Part B: bupivacaine HCl (Active Comparator): Children ≥6 to <12 years of age. A single dose of bupivacaine HCl 0.25% (without epinephrine) via injection into the surgical site
  Interventions: Drug: Bupivacaine HCl
- Cohort 3: HTX-011 (Experimental): Children ≥3 to <6 years of age. Dose to be determined from Cohorts 1 and 2.
  Interventions: Drug: HTX-011; Device: Luer Lock Applicator
- Cohort 3: bupivacaine HCl (Active Comparator): Children ≥3 to <6 years of age. A single dose of bupivacaine HCl 0.25% (without epinephrine) via injection into the surgical site
  Interventions: Drug: Bupivacaine HCl

INTERVENTIONS:
Drug: HTX-011 — Single-dose instillation of approximately 0.17 mL/kg (total dose does not exceed 10.5 mL) of HTX-011.
  Arms: Cohort 1 Part A: HTX-011
Drug: Bupivacaine HCl — Bupivacaine HCl 0.25% (without epinephrine) (total dose not to exceed 75 mg).
  Arms: Cohort 1 Part A: bupivacaine HCl; Cohort 1 Part B: bupivacaine HCl; Cohort 2 Part A: bupivacaine HCl; Cohort 2 Part B: bupivacaine HCl; Cohort 3: bupivacaine HCl
Drug: HTX-011 — Dose to be determined from Cohort 1.
  Arms: Cohort 2 Part A: HTX-011; Cohort 2 Part B: HTX-011
Drug: HTX-011 — Dose to be determined from Cohorts 1 and 2.
  Arms: Cohort 3: HTX-011
Drug: HTX-011 — Dose to be determined from Cohort 1 Part A.
  Arms: Cohort 1 Part B: HTX-011
Device: Luer Lock Applicator — Applicator for instillation.
  Arms: Cohort 1 Part A: HTX-011; Cohort 1 Part B: HTX-011; Cohort 2 Part A: HTX-011; Cohort 2 Part B: HTX-011; Cohort 3: HTX-011

SUMMARY:
This is a Phase 2 study in pediatric subjects undergoing inguinal herniorrhaphy.

ELIGIBILITY:
Inclusion Criteria:

* Is scheduled to undergo a unilateral open inguinal herniorrhaphy with or without mesh under general anesthesia.
* Has an American Society of Anesthesiologists Physical Status of I, II, or III.
* Female subjects are eligible only if not pregnant, not lactating, not planning to become pregnant during the study, sterile; or using acceptable contraceptives.

Exclusion Criteria:

* Has a medical condition such that, in the opinion of the Investigator, participating in the study would pose a health risk to the subject or confound the postoperative assessments.
* Has a planned concurrent surgical procedure (eg, bilateral herniorrhaphy).
* Has a contraindication or a known or suspected history of hypersensitivity or clinically significant idiosyncratic reaction to required study medications.
* Has taken meloxicam within least 10 days prior to the scheduled surgery.
* Has been administered bupivacaine within 5 days prior to the scheduled surgery.
* Has been administered any local anesthetic within 72 hours prior to the scheduled surgery.
* Has a known or suspected history of drug abuse, a positive drug screen on the day of surgery, or a recent history of alcohol abuse. Note: Subjects with a positive drug screen who are taking an allowed, prescribed medication that is known to result in a positive drug test (eg, amphetamine and dextroamphetamine for attention-deficit/hyperactivity disorder, benzodiazepine for anxiety disorder) may be eligible for participation in the study at the discretion of the Sponsor. Subjects taking any marijuana (medical or recreational) are not allowed to participate in the study.
* Previously participated in an HTX-011 study.
* Received an investigational product or device in a clinical trial within 30 days or within 5 elimination half-lives.
* Has a body mass index (BMI) >35 kg/m2.

In addition to the preceding exclusion criteria 1 through 14, subjects to be enrolled in Cohort 1 Part B, Cohort 2 Part B, or Cohort 3 who meet any of the following criteria prior to randomization will be excluded from the study:

* Has had a prior ipsilateral inguinal herniorrhaphy.
* Has a pre-existing concurrent acute or chronic painful physical/restrictive condition expected to require analgesic treatment in the postoperative period for pain.
* Has known or suspected daily use of opioids for 7 or more consecutive days within the previous 6 months.
* Has taken long-acting opioids within 3 days prior to the scheduled surgery.
* Has taken any opioids within 48 hours prior to the scheduled surgery.
* Has initiated treatment with study medications within 1 month prior to study drug administration that can impact pain control.
* Has been administered systemic steroids within 5 half-lives or 10 days prior to administration of study drug.
* Has undergone 3 or more surgeries within 12 months.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) from Time 0 extrapolated to infinity (AUCinf) | 72 hours
Maximum concentration (Cmax) | 72 hours
Time of occurrence of maximum concentration (Tmax) | 72 hours

SECONDARY OUTCOMES:
Adolescents ≥12 to <17 years of age (Cohort 1): area under the curve (AUC) of the Numeric Rating Scale of pain intensity scores with activity (NRS-A) | 72 hours
Children ≥6 to <12 years of age (Cohort 2): AUC of the Faces-Pain-Scale (FPS)-Revised pain intensity scores | 72 hours
Children ≥3 to <6 years of age (Cohort 3): AUC of the Faces, Legs, Activity, Cry, Consolability (FLACC) scale pain intensity scores | 72 hours
Total postoperative opioid consumption (in IV morphine milligram equivalents) | 72 hours
Proportion of subjects who are opioid-free | 72 hours
AUC of the Numeric Rating Scale pain intensity scores at rest (NRS-R) | 72 hours
Proportion of subjects who do not receive an opioid prescription at discharge. | 72 hours

IPD SHARING:
Plan to Share IPD: Undecided